CLINICAL TRIAL: NCT06111976
Title: Repetitive Transcranial Magnetic Stimulation Plus Reactivation Therapy Efficacy on PTSD Symptom Severity in Resistant PTSD, a Randomized Double Blind Sham Controlled Trial (TraumaStim)
Brief Title: Repetitive Transcranial Magnetic Stimulation Plus Reactivation Therapy Efficacy on PTSD Symptom Severity in Resistant PTSD
Acronym: TraumaStim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP200044; 2021-A02532-39-B (Other: IDRCB ANSM)
Record Dates: First submitted 2023-10-12; First posted 2023-11-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Stress Disorders; Traumatic Stress Disorders; Post-Traumatic Trauma and Stressor Related Disorders; Mental Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Mental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS with simultaneous reactivation of traumatic memory in resistant PTSD (Experimental): rTMS with simultaneous reactivation of traumatic memory in resistant PTSD during 12 sessions (3 to 4 weeks)
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)
- sham rTMS and simultaneous reactivation of traumatic memory in resistant PTSD (Placebo Comparator): sham rTMS and simultaneous reactivation of traumatic memory in resistant PTSD during 12 sessions (3 to 4 weeks)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS with simultaneous reactivation of traumatic memory will be performed 3 to 4 times a week for 3 to 4 weeks through 12 sessions.
  A traumatic script will be prepared by the patient at the inclusion visit, which will be used to reactivate the traumatic memory after every rTMS or sham rTMS sessions.
  Arms: rTMS with simultaneous reactivation of traumatic memory in resistant PTSD
Procedure: Placebo — sham rTMS with simultaneous reactivation of traumatic memory will be performed 3 to 4 times a week for 3 to 4 weeks through 12 sessions.
  A traumatic script will be prepared by the patient at the inclusion visit, which will be used to reactivate the traumatic memory after every rTMS or sham rTMS sessions.
  Arms: sham rTMS and simultaneous reactivation of traumatic memory in resistant PTSD

SUMMARY:
A French multicenter randomized and double blinded shamed controlled study recruiting patients who present resistant PTSD. The aim of this trial is to assess the efficacy of cerebral modulation by rTMS with simultaneous reactivation of traumatic memory on the PTSD symptoms at M1.

DETAILED DESCRIPTION:
Detailed Description : PTSD is considered as one of the top 10 public health concerns. Most patients with PTSD receive pharmacologic treatment and traumatic reactivation therapy. However, to date, the optimal treatment alternatives for non-responders PTSD patients are unknown.

Functionally, the metabolic activity of the prefrontal-amygdala cortex circuit in PTSD is significantly altered. Repetitive Transcranial Magnetic Stimulation (rTMS) provides focused, non-invasive stimulation of cortical areas of the central nervous system and could correct cortical defective activation of the prefrontal cortex seen in PTSD Patient (FDA has already approved rTMS for depression and acoustic-verbal hallucinations treatment).

Pairing rTMS with cues relevant to the trauma may be a novel approach to treat PTSD patient.

The study will enroll 102 subjects with resistant PTSD. After screening and inclusion phase, the treatment phase with 12 sessions of rTMS and simultaneous reactivation of traumatic memory or sham rTMS and simultaneous reactivation of traumatic memory will be performed (3 to 4 weeks). Antidepressant treatment will be maintained. The follow up phase consist of 3 visits at M1, M3 and M6 to follow the evolution of the PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years.
* Presenting a PTSD according to DSM-5 criteria
* Patient with persistent symptoms (PCL-5>40) after a 6 weeks treatment with labelled antidepressant for PTSD (paroxetine or sertraline)
* Patient with health insurance (AME excepted)
* Signed written inform consent

Exclusion Criteria :

* Contraindication for rTMS:

  * History of epilepsy or seizure
  * Cochlear implants
  * Cardiac pacemaker or intracardiac lines, or metal in the body
* Patient has already had a rTMS session and/or Electroconvulsive therapy (ECT) and/or Transcranial direct current stimulation (tDCS)
* Ongoing PTSD-oriented cognitive-behavioral therapy
* Lifetime psychotic or bipolar disorder or antisocial personality or borderline personality
* Brain injury defined by medical report (including cortical and subcortical atrophy, dementia, stroke, transient ischemic attack and head trauma)
* Current substance dependence (including alcohol, excluding tobacco);
* Acute suicidal ideation
* No adequate mastering of the French language or no ability to consent
* Pregnancy (confirmed by a urine test beta-HCG) or breast feeding or absence of birth control
* Patient under legal protection measure and or deprived of freedom
* Participation in any other interventional study or in the exclusion period any other interventional study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
PTSD severity score measured at M1 after 12 sessions of rTMS or sham rTMS and simultaneous reactivation of traumatic memory | Month 1 after 12 sessions of rTMS
  CAPS-5 total severity score at M1 post treatment will be compared between groups (cerebral modulation by rTMS with simultaneous reactivation of traumatic memory VS sham rTMS with simultaneous reactivation of traumatic memory)

SECONDARY OUTCOMES:
PTSD severity scores at M3 and M6 measured with CAPS-5 | At inclusion (v1), Month 3 and Month 6 post treatment
  The different dimensions of PTSD (assess by CAPS-5): Severity, repetition, avoidance, neurovegetative activation at M3 and M6 post treatment
The severity of PTSD assessed by PCL-5 at each visit. | at once a during TMS sessions, Month1, Month 3 and Month 6 post treatment.
  PTSD severity score measured with the PTSD Checklist (PCL-S self-questionnaire) at once a during TMS sessions, M1, M3 and M6 post treatment
Dissociative symptoms severity scores (1) | at inclusion (V1), up to 4 weeks (V13) (end of treatment), Month 1, Month 3, Month 6 post treatment
  Dissociative symptoms severity score measured with the Clinician Administered Dissociative States Scale (CADSS)
Dissociative symptoms severity scores (2) | at inclusion (V1), up to 4 weeks (V13) (end of treatment), Month 1, Month 3, Month 6 post treatment
  The Multidimensional Assessment of Interoceptive Awareness (MAIA)
Dissociative symptoms severity scores (3) | at inclusion (V1), up to 4 weeks (V13) (end of treatment), Month 1, Month 3, Month 6 post treatment
  The Dissociative Experiences Scale (DES)
The severity scores of the dimensions of anxiety at V13 (end of treatment), M1, M3, M6 post treatment. | Up to 4 weeks (V13) (end of treatment), Month 1, Month 3, Month 6 post treatment.
  The severity scores of the dimensions of anxiety measured with HAM-A at V13 (end of treatment), M1, M3 and M6.
Symptoms of depression at V13 (end of treatment), M1, M3, M6 post treatment. | at V13 (end of treatment), Month 1, Month 3, Month 6 post treatment.
  The severity scores of the dimensions of depression measured with HAM-D at V13 (end of treatment), M1, M3 and M6.
Evolution of social cognition at M3 post treatment. | at Month 3 post treatment
  Evolution of social cognition at M3 post treatment by a neuropsychologist
Quality of life | post treatment and Month 6
  Quality of life evolution post treatment and M6 assessed by WHOQOL EuroQol Health Measure
Quality of life | post treatment and Month 6
  Quality of life evolution post treatment and M6 assessed by EQ-5D-5L
Proportion of adverse events during the active treatment phase and during the follow-up | through study completion, up to 6 months
  Number and description of adverse events during the active treatment phase and during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Florian FERRERI, MD, ph, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital, Psychiatry department, Assistance Publique- Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No